CLINICAL TRIAL: NCT05983640
Title: Just in Time Cardio Pulmonary Resuscitation Trial (JITCPR-T): Comparison of a Brief Video to Traditional CPR Training: a Randomized Controlled Trial
Brief Title: Just in Time Cardio Pulmonary Resuscitation Trial
Acronym: JITCPR-T
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Massachusetts General Hospital (Other); American Heart Association (Other)
Responsible Party: Principal Investigator, Eric Goralnick, Associate Professor of Emergency Medicine, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2023P000222
Record Dates: First submitted 2023-04-12; First posted 2023-08-09 (Actual); Last update posted 2023-08-09 (Actual); Status verified 2023-08

CONDITIONS: Cardiopulmonary Arrest With Successful Resuscitation; Educational Problems
Keywords: Youtube; Video Education; Public Empowerment; CPR; AED
MeSH Terms: interventions — Videotape Recording

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, three arm, parallel, open-label trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention): Assessment without training or video prompt
- Just in time video (Experimental): Assessment with JiT video available
  Interventions: Other: Video
- AHA Course (Active Comparator): Assessment after completion of CPR training course
  Interventions: Other: AHA course

INTERVENTIONS:
Other: Video — Just in time training video on hands only CPR
  Arms: Just in time video
Other: AHA course — AHA Heartsaver CPR course
  Arms: AHA Course

SUMMARY:
The objective is to evaluate the effectiveness of a Just in Time (JiT) video as compared to the AHA Heartsaver® Course and no training (control) in ability to correctly perform CPR. The secondary objective is to assess skill retention 3-9 months after the AHA Heartsaver course with and without JiT Video use. The goal of this work is to study the effectiveness of this new JiT video to improve objective knowledge- and performance-based measures of effective OHCA response, as well as subjective ratings of preparedness and likeliness to respond, compared to the standard AHA Heartsaver® CPR AED Training course.

DETAILED DESCRIPTION:
The first responder phase of out-of-hospital cardiac arrest (OHCA) response is most often led by bystanders with limited resources and no medical training. Bystanders play a critical role in the initial measures of the cardiac arrest chain of survival-activation of emergency medical services (EMS), initiation of cardiopulmonary resuscitation (CPR), and administration of defibrillation when indicated. Early bystander response, early bystander CPR, and defibrillation in under 8 minutes are associated with increased survival to hospital discharge.

Despite the clear importance of early bystander response to OHCA, rates of bystander CPR remain low with only one-third of OHCA patients receiving bystander CPR. Lay people with CPR training are more likely to perform CPR than those without training. Prior studies comparing traditional in-person training programs for CPR versus technology-enabled self-instruction (TESI) formats have demonstrated superiority or equivalency of TESI to prepare lay bystanders in OHCA response. Shorter duration and more convenient access to TESI in light of these findings provide a promising opportunity to increase public preparedness to participate in OHCA management at greater scales and lower costs. However, CPR-specific skills and knowledge deteriorate within 3 to 6 months of initial training, and time, location, and duration have all been perceived as barriers to completing CPR training.

The objective is to evaluate the effectiveness of a Just in Time (JiT) video as compared to the AHA Heartsaver® CPR AED Training Course and no training (control) in ability to correctly perform CPR. The secondary objectives are the evaluation participate interaction with the JiT video and to assess skill retention 3-9 months after the AHA Heartsaver course with and without JiT Video use. The goal of this work is to study the effectiveness of this new JiT video to improve objective knowledge- and performance-based measures of effective OHCA response, as well as subjective ratings of preparedness and likeliness to respond, compared to the standard AHA Heartsaver® CPR AED Training course.

This is a prospective, randomized, three arm, open-label trial will two rounds of data collection. In the first round, participants will be randomized to one of three arms (no training, AHA course, JiT video) and assessed on CPR skills and knowledge. All participants will then be exposed to the other conditions (completion of the AHA Heartsaver® CPR AED Training course and viewing of the JiT video). During the second round, approximately 3-12 months later, the investigators will test the effectiveness of the JiT video at prompting correct CPR skills after previous training versus no prompting.

Specific aim 1: Determine the efficacy of an abbreviated JiT video-based curriculum in achieving competence in CPR by lay-persons as compared to individuals trained by the AHA Heartsaver® CPR AED Training course.

Hypothesis 1: Participants in the abbreviated JiT video-based curriculum will have no difference in measures of objective knowledge, objective performance, and subjective preparedness to administer CPR compared to participants in the in-person AHA Heartsaver® CPR AED Training course, but superior results compared to controls.

Specific aim 2: Determine how participants interact with a JiT CPR education video during a simulated cardiac arrest. This is an exploratory, qualitative aim.

Specific aim 3: Determine retention of CPR skills using the abbreviated JiT video between 3-12 months after initial training, as compared to retention from the AHA Heartsaver® CPR AED Training course alone without a refresher.

Hypothesis 3: Participants who view the abbreviated JiT video during reassessment will have no differences in measures of objective knowledge, objective performance, and subjective preparedness to administer CPR compared to those without the video 3-12 months after initial training, but superior results compared to controls.

ELIGIBILITY:
Inclusion Criteria:

* Employee of Gillette Stadium

Exclusion Criteria:

* Age less than 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2023-03-27 (Actual); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-01-01 (Estimated)

PRIMARY OUTCOMES:
Performance of correct cardiopulmonary resuscitation (CPR) (Objective Performance) | Measured within 2 hours of randomization, during the intervention
  Correct CPR will be measured by successful completion of all five of the following actions:
  1. Calling for 9-1-1 (as measured by verbalizing action to examiner)
  2. Calling for automated external defibrillator (as measured by verbalizing action to examiner)
  3. Placing hand in correct position on manikin chest (as measured by examiner)
  4. Compressing at a rate of 100-120 per minute (as measured by examiner and through CPR manikin equipped with Laerdal QCPR software)
  5. Compressing to a depth of at least 2 inches (as measured by examiner and through CPR manikin equipped with Laerdal QCPR software)

SECONDARY OUTCOMES:
CPR knowledge (Objective Knowledge) | Measured immediately after skill evaluation completion
  Knowledge regarding CPR skills will be measured by an 8-question multiple choice assessment, based on the American Heart Association HeartSaver curriculum. The assessment will test participants' understanding of when to perform CPR on a victim and how to perform CPR correctly (e.g., hand placement, compression rate, and compression depth). The assessment will be scored as 1 point per correct answer, with a range of 0-8 points (higher score indicates better knowledge).
Change in willingness to respond (Subjective Preparedness) | Measured within 1 hour before and immediately after skill evaluation completion
  Participants will complete pre/post 6-question assessments to determine the change in their likelihood and confidence in providing CPR in different situations. Items will be scored on a 5-point Likert-type scale (very unlikely to very likely) for likelihood to perform CPR (for a stranger, close relative for friend, or if requested by a trained professional and confidence in identifying cardiac arrest, performing CPR, and using an AED. Change in willingness to respond will be measured by examining the within-person change from pre and post assessments.

CONTACTS AND LOCATIONS:
Overall Officials: Eric Goralnick, MD, MS, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Gillette Stadium, Foxborough, Massachusetts, United States

REFERENCES:
- [Derived] Goldberg SA, Cash RE, Peters GA, Jiang D, O'Brien C, Hasdianda MA, Eberl EM, Salerno KJ, Lees J, Kaithamattam J, Tom J, Panchal AR, Goralnick E. Evaluating video-supported layperson CPR compared to a standard training course: A randomized controlled trial. Resusc Plus. 2024 Dec 6;20:100835. doi: 10.1016/j.resplu.2024.100835. eCollection 2024 Dec. PMID 39717499